CLINICAL TRIAL: NCT05513989
Title: Modified Magill Forceps Facilitating Nasal Intubation for Children Undergoing Dental Operations
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, RAMY AHMED, Assistant Professor of Anesthesia, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IRB00006379 MMF
Record Dates: First submitted 2022-08-16; First posted 2022-08-24 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Endotracheal Tube Wrongly Placed During Anesthetic Procedure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- modified Magill forceps group (Active Comparator): One hundred and ten patients for whom modified pediatric Magill forceps was used to assist nasotracheal intubation
  Interventions: Device: modified Magill forceps
- Magill forceps group (Active Comparator): One hundred and ten patients for whom Magill forceps was used to assist nasotracheal intubation.
  Interventions: Device: Magill forceps

INTERVENTIONS:
Device: modified Magill forceps — modified pediatric Magill forceps was used to assist nasotracheal intubation.
  Arms: modified Magill forceps group
Device: Magill forceps — Magill forceps was used to assist nasotracheal intubation.
  Arms: Magill forceps group

SUMMARY:
compare between Magill forceps and modified pediatric Magill forceps for nasotracheal intubation (which method is easier and better?).

DETAILED DESCRIPTION:
Group A One hundred and ten patients for whom modified pediatric Magill forceps was used to assist nasotracheal intubation.

Group B One hundred and ten patients for whom Magill forceps was used to assist nasotracheal intubation.

For each patient, intubation time, number of intubation attempts, hypoxia (recognized when oxygen saturation decreases below 94%), pharyngeal trauma, and need for corkscrewing will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the American Society of Anesthesiology physical status of 1 or 2
* Age 4 to 8 years old.
* Elective dental surgeries.

Exclusion Criteria:

* Parental refusal to consent (absolute contraindication),
* Patients with aspiration risk.
* Known upper airway abnormalities.
* Those having difficult airway.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
intubation time | just after anesthesia induction for 30 minutes

SECONDARY OUTCOMES:
number of intubation attempts | after anesthesia induction for 30 minutes
hypoxia | after anesthesia induction for 30 minutes
pharyngeal trauma | after intubation for 30 minutes
need for corkscrewing | after anesthesia induction for 30 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Ain shams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No